CLINICAL TRIAL: NCT00004172
Title: Peripheral Stem Cell Transplantation Protocol for Patients With Previously Treated Advanced Breast Cancer - A Phase II Pilot Study
Brief Title: Chemotherapy, Filgrastim, and Stem Cell Transplantation With Radiation Therapy in Treating Patients With Stage III or Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 92B3T; NU-92B3T; NCI-G99-1640
Record Dates: First submitted 1999-12-10; First posted 2004-09-16 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Ifosfamide; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: ifosfamide
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. Combining chemotherapy with autologous peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to compare the effectiveness of two regimens of chemotherapy and filgrastim plus stem cell transplantation in treating patients who have previously untreated stage III or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor response, survival, and disease free survival following high dose carboplatin, ifosfamide, and thiotepa with autologous peripheral blood stem cell (PBSC) support and consolidation radiotherapy to sites of pretreatment bulk disease in patients with previously treated advanced breast cancer. II. Assess the toxicity of high dose chemotherapy in these patients. III. Compare the effectiveness of PBSC mobilization with high dose cyclophosphamide and filgrastim (G-CSF) vs G-CSF alone in this patient population.

OUTLINE: Patients are assigned to 1 of 2 peripheral blood stem cell (PBSC) mobilization groups at the discretion of the attending physician: Group 1: Patients receive high dose cyclophosphamide IV over 6 hours and filgrastim (G-CSF) subcutaneously (SQ) daily beginning 24 hours after completion of cyclophosphamide and continuing until 3 days after blood counts have recovered and until PBSC are harvested. Group 2: Patients receive G-CSF SQ daily alone until PBSC are harvested. Both groups: PBSC are harvested on days 15-19 after cyclophosphamide infusion or when blood counts recover. Patients receive high dose carboplatin IV continuously, ifosfamide IV over 4 hours, and thiotepa IV over 1 hour on days -5 to -3. PBSC are reinfused beginning 48 hours after completion of combination chemotherapy. Patients receive G-CSF SQ beginning on day 0 and continuing until 3 days after blood counts have recovered. Sites of pretransplantation metastases greater than 3 cm are irradiated beginning after transplantation and after blood counts recover. Patients are followed every month for 1 year.

PROJECTED ACCRUAL: A total of 12-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven previously treated stage III or IV breast cancer No CNS disease Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Physiologic 65 and under Menopausal status: Not specified Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Hepatic function normal unless due to liver metastases Bilirubin less than 1.5 times normal SGOT or SGPT less than 1.5 times normal Alkaline phosphatase less than 1.5 times normal If hepatitis C antibody positive, then liver function must be normal OR liver dysfunction must be due to metastatic disease and not chronic hepatitis Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: LVEF normal No myocardial infarction within past 6 months No significant arrhythmia requiring medications No history of congestive heart failure Pulmonary: DLCO at least 50% predicted FEV1 and/or FVC at least 75% predicted No serious nonneoplastic pulmonary disease (severe chronic obstructive lung disease) that would preclude study therapy Other: Not pregnant Negative pregnancy test HIV negative Hepatitis B and C surface antigen negative No active serious medical condition that would preclude study therapy

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane N. Winter, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States